CLINICAL TRIAL: NCT07401108
Title: Reactive Balance Training Versus Virtual Reality on Balance and Functional Abilities in Children With Hemiplegia
Brief Title: Reactive Balance Training vs Virtual Reality in Hemiplegic Cerebral Palsy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Esraa Abd Elaziz Anter, lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/005531
Record Dates: First submitted 2026-01-05; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Hemiplegic Cerebral Palsy
Keywords: Virtual Reality; Hemiplegic Cerebral Palsy; Wii Balance Board; Reactive Balance Training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality using Wii Balance Board (Experimental): The Wii Balance Board is a non-immersive virtual reality (VR) rehabilitation tool that has been widely used in physical therapy to assess and train balance and postural control. It is a force-platform-based device equipped with four pressure sensors (anterior-posterior and medial-lateral) that detect changes in body weight distribution and shifts in the center of pressure (CoP). These data are transmitted in real time to the Nintendo Wii console, where body movements are translated into visual feedback displayed on a screen, allowing users to interact with virtual environments and game-based tasks.
  Interventions: Device: Virtual reality
- Reactive Balance training (Experimental): Participants will undergo structured reactive balance training that will consist of three sessions per week over an eight-week period. In Reactive balance training we will use different types of perturbations: External perturbations, Internal perturbation and combination of them. Training will last about 30 minutes.
  Interventions: Other: Reactive Balance Training

INTERVENTIONS:
Device: Virtual reality — Participants will undergo a structured balance training program utilizing the Wii Balance Board. The program will consist of three training sessions per week over an eight-week period.
  The first two weeks will focus on guided exercises with manual assistance and verbal instructions, ensuring that the children are comfortable and correctly performing the exercises. As the participants progress, the manual guidance will be gradually reduced, and verbal instructions alone will be provided for the remaining four weeks of training.
  Other Names: Wii Balance Board
  Arms: Virtual reality using Wii Balance Board
Other: Reactive Balance Training — In reactive balance training, each session will include 3-4 of the following five core exercises: lean and release, push/pull, reaching with unexpected perturbation, weight shifting on unstable surfaces, and trip/slip simulation. Exercises will be divided into 2-3 blocks, with 6-8 perturbations in each block and short rest periods between blocks (1-2 min), for a total of 30-40 perturbations per session.
  Other Names: Perturbation- Based Training
  Arms: Reactive Balance training

SUMMARY:
This randomized controlled study compared the effects of Wii Balance Board training versus reactive balance training on balance control and functional abilities in children with spastic hemiplegic cerebral palsy. Sixty children aged 6-10 years (GMFCS levels I-II, mild spasticity) were randomly assigned to either a Wii-based balance training group or a reactive balance training group. Both groups received a conventional physical therapy program three times per week for eight weeks, with an additional 30 minutes of the assigned balance intervention per session. Balance and functional abilities were assessed before and after treatment using the HUMAC Balance System, Pediatric Balance Scale, Functional Reach Test, and Timed Up and Down Stairs test. The study aimed to evaluate and compare the effectiveness of both interventions in improving balance control and functional performance in this population.

DETAILED DESCRIPTION:
This study was conducted as a randomized controlled trial to investigate and compare the effects of Wii Balance Board-based virtual reality training and reactive balance training on balance control and functional abilities in children with spastic hemiplegic cerebral palsy.

Study Design and Participants

Sixty children with spastic hemiplegia of both genders were recruited from Wahet Nour Elhayah Centers. Participants were aged between 6 and 10 years, classified as GMFCS levels I and II, and demonstrated mild spasticity (grades 1-1+ on the Modified Ashworth Scale). All children were able to follow verbal instructions and participate actively in assessment and treatment procedures. Children with musculoskeletal deformities, recent orthopedic surgery or botulinum toxin injections, uncontrolled seizures, cardiovascular or respiratory disorders, or visual or hearing impairments were excluded.

Participants were randomly allocated into two equal groups (Group A and Group B) using a simple randomization method.

Intervention Program

Both groups received a conventional physical therapy program for 90 minutes per session, three times per week for eight weeks. This program included neurodevelopmental treatment techniques, stretching exercises for affected upper and lower limbs, upper limb strengthening and functional exercises, and gait training.

In addition to conventional therapy, each group received a specific balance training intervention for 30 minutes per session.

Group A: Wii Balance Board Training (Virtual Reality-Based Balance Training)

Children in Group A participated in a structured balance training program using the Nintendo Wii Balance Board. Training was conducted three times per week for eight weeks. The program was designed to improve static and dynamic balance, weight-shifting ability, and sensorimotor integration through interactive virtual reality games.

During the first two weeks, training focused on familiarization with the device and games, with close therapist supervision, manual assistance, and verbal cues to ensure proper movement execution and safety. As participants progressed, manual assistance was gradually withdrawn, and training during the remaining weeks relied primarily on verbal instructions.

Each session was divided into three series. The first and second series included games such as Snowboard, Penguin Slide, and Super Hula Hoop, which required continuous weight shifting in the anteroposterior, mediolateral, and combined directions. Short rest periods (1-2 minutes) were provided between series to prevent fatigue. The third series involved relaxation and postural control exercises using the Yoga game, initially performed with eyes open and later with eyes closed to challenge sensory integration.

This training approach emphasized continuous visual feedback, motivation, and active participation, aiming to enhance postural control through multisensory stimulation and task-oriented practice.

Group B: Reactive Balance Training

Children in Group B received a structured reactive balance training program, also delivered three times per week for eight weeks, with each session lasting approximately 30 minutes. The goal of this intervention was to improve the child's ability to recover balance in response to unexpected perturbations.

Training included external perturbations, internal perturbations, and combinations of both. External perturbations were applied by the therapist through techniques such as lean-and-release maneuvers and sudden, unpredictable pushes to the shoulder or pelvis while the child stood on a stable or unstable surface. Children were instructed to maintain balance with minimal displacement of the center of gravity. Internal perturbations involved voluntary destabilizing tasks such as kicking or throwing a ball while maintaining postural stability.

As participants' reactive balance responses improved, task difficulty was progressively increased by modifying perturbation magnitude, direction, and unpredictability, as well as by introducing sensory challenges or unstable support surfaces. This progression aimed to simulate real-life balance disturbances and enhance rapid postural responses.

Outcome Measures and Assessment Procedures

All participants were evaluated before and after the 8-week intervention period. Balance was objectively assessed using the HUMAC Balance System, including measures of center of pressure, limits of stability, and weight-shifting ability. Functional balance was assessed using the Pediatric Balance Scale. Functional performance was evaluated using the Functional Reach Test and the Timed Up and Down Stairs (TUDS) test.

Purpose of the Protocol

This protocol was designed to determine the effectiveness of Wii-based virtual reality training and reactive balance training in improving balance control and functional abilities in children with spastic hemiplegia, and to compare which approach yields superior clinical outcomes. The results are intended to guide evidence-based balance rehabilitation strategies for this population.

ELIGIBILITY:
Inclusion Criteria:

* Hemiplegic children between 6-10 years old.
* Both genders will be included.
* Their motor function will be between level I and II according to Gross Motor Function Classification System (GMFCS) .
* The degree of spasticity for these children will range from grade 1 to 1+ according to the Modified Ashworth Scale .
* They will be able to follow instructions during evaluation and treatment procedures

Exclusion Criteria:

* Cardiovascular or respiratory disorders.
* Undergone musculoskeletal surgery or botulinum toxin injection in the lower limbs in past six months
* Musculoskeletal problems or fixed deformities in the spine and/or lower extremities
* unstable seizures
* Visual or hearing impairment

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2025-05-24 (Actual); Primary Completion 2026-02-23 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Limits of stability scores | From enrollment to the end of treatment at 8 weeks
  The Humac Balance System will be used for assessment of balance through limits of stability (LOS) scores. Higher scores indicate better dynamic balance control
center of pressure scores | From enrollment to the end of treatment at 8 weeks
  The Humac Balance System will be used for assessment of balance through center of pressure (COP) scores. Lower values indicate better posture control

SECONDARY OUTCOMES:
Functional reach test scores | From enrollment to the end of treatment at 8 weeks
  Functional abilities will be assessed using the functional reach test measured in centimeters. Higher reach distance indicates better functional balance
Timed up-and-down-stairs test scores | From enrollment to the end of treatment at 8 weeks
  Functional abilities will be assessed using timed up and down stairs measured in seconds. Lower time indicates better functional performance

CONTACTS AND LOCATIONS:
Locations (1):
- Wahet nour elahayah, Al Mansurah, Daqahlyia, Egypt